CLINICAL TRIAL: NCT00430911
Title: Radiotherapy for Malignant Astrocytomas in the Elderly
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC, P000502 AOM 98071
Record Dates: First submitted 2007-01-31; First posted 2007-02-02 (Estimated); Last update posted 2007-02-02 (Estimated); Status verified 2007-01

CONDITIONS: Primary Brain Tumor; Anaplastic Astrocytoma; Glioblastoma Multiforme
Keywords: malignant gliomas
MeSH Terms: conditions — Brain Neoplasms; Astrocytoma; Glioblastoma; Glioma | interventions — Radiotherapy

INTERVENTIONS:
Drug: Radiotherapy

SUMMARY:
A randomized trial comparing radiotherapy with supportive care in patients aged 70 years or older with newly diagnosed, histologically confirmed anaplastic astrocytoma or glioblastoma, and a Karnofsky performance status > 70.

ELIGIBILITY:
Inclusion Criteria:

* Glioblastoma and anaplastic astrocytoma, supratentorial, histologically confirmed
* Brain CT scan or MRI within 28 days before surgery
* Age: 70 years or older
* Karnofsky performance status, 70 or more.
* Life expectancy over 12 weeks
* Informed consent

Exclusion Criteria:

* Brain radiotherapy
* Chemotherapy
* Severe systemic disease

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Dates: Start 2001-02

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
Progression free survival
Quality of life
Cognitive functions

CONTACTS AND LOCATIONS:
Overall Officials: jean-yves Delattre, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Florence Keime-Guibert, MD, Principal Investigator — Assitance Publique-Hôpitaux de Paris
Locations (1):
- Hôpital de la Salpêtrière, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Keime-Guibert F, Chinot O, Taillandier L, Cartalat-Carel S, Frenay M, Kantor G, Guillamo JS, Jadaud E, Colin P, Bondiau PY, Menei P, Loiseau H, Bernier V, Honnorat J, Barrie M, Mokhtari K, Mazeron JJ, Bissery A, Delattre JY; Association of French-Speaking Neuro-Oncologists. Radiotherapy for glioblastoma in the elderly. N Engl J Med. 2007 Apr 12;356(15):1527-35. doi: 10.1056/NEJMoa065901. PMID 17429084